CLINICAL TRIAL: NCT01203839
Title: A Phase II Study of Partial Breast Irradiation (PBI) Using 40 Gy for Select Patients With Early Invasive or Noninvasive Breast Cancer
Brief Title: Partial Breast Irradiation (PBI) Using 40 Gy for Select Patients With Early Invasive or Noninvasive Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-114
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: stage 1 breast cancer; invasive ductal breast; Partial Breast Irradiation (PBI); radiation; 10-114
MeSH Terms: conditions — Breast Neoplasms

ARMS (1):
- Radiation treatment (Experimental): This is a Phase II single-arm study of PBI with external-beam radiation therapy in which a group of select women with early-stage invasive and noninvasive breast cancer will be given radiation to the partial breast.
  Interventions: Radiation: multiple beams utilizing either intensity-modulated or 3D-conformal techniques

INTERVENTIONS:
Radiation: multiple beams utilizing either intensity-modulated or 3D-conformal techniques — A dose of 40 Gy will be delivered to the tumor bed plus 1.5-2 cm margin. Treatment will be delivered once daily, 5 days a week, for approximately 2 weeks. Radiation therapy will begin within a minimum of 4 weeks and a maximum of 3 months from definitive surgical procedure and 2-6 weeks after chemotherapy, if chemotherapy given first. Prior to radiation, patients will receive a lumpectomy with an assessment of axillary lymph node status (for invasive tumors only). Axillary assessment may be any combination of sentinel lymph node biopsy or axillary lymph node dissection.

SUMMARY:
Currently the standard of care is to treat early stage invasive breast cancer or ductal carcinoma in situ (DCIS) with a combination of lumpectomy and radiotherapy, known as "breast-conserving therapy" (BCT). The traditional method of giving radiation therapy after a lumpectomy is to the whole breast.

However the investigators do not know if the whole breast needs to be receive radiation to better control your cancer or only a more limited area of the breast surrounding the tumor. The purpose of this study is to see the side effects of delivering partial breast irradiation (PBI) instead of whole breast irradiation (WBI). PBI is radiation therapy given only to the area of the breast where the cancer was removed. Another purpose of this study is to look long term at the rate at which cancer comes back in the same breast after PBI.

WBI is radiation therapy given 5 days a week for 5 to 7 weeks to the whole breast. Partial breast irradiation radiation therapy (PBI) is much shorter than whole breast irradiation. The investigators propose to deliver the PBI radiation therapy, for a few minutes a day, once a day, five days a week, for 2 weeks.

In this study the investigators will learn about the good and bad effects of PBI radiation therapy. In this study, the investigators will also learn about how the breast looks after surgery and radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age ≥ 18 years
* Unicentric Stage I (T1N0M0) invasive ductal breast cancer or Grade 1 or II DCIS measuring <2 cm on pathology and/or mammogram that is histologically confirmed at MSKCC
* Histologically negative tumor margin 2 mm or more from any inked edges or no tumor in a re-excision specimen or final shaved specimen
* ECOG Performance Status of 0 or 1
* Granulocytes ≥1,500/μl and platelet count must be ≥100,000/μl at the beginning of therapy for patients treated with adjuvant chemotherapy
* Women >70 years or older with T1 invasive ductal carcinoma who are estrogen-receptor positive (ER+) with clinically negative axillary nodes and do not undergo surgical lymph node evaluation are eligible if patient will take hormonal therapy.
* Patients with T1N0(i+) tumors on sentinel lymph node mapping or dissection (i.e., if tumor deposit is 0.2 mm or less, regardless of whether the deposit is detected by immunohistochemistry or hematoxylin and eosin staining) will also be eligible.
* Clips must be placed in the lumpectomy cavity at the time of final excision in order to aid in the delineation of the tumor cavity at the time of simulation and radiation delivery.

Exclusion Criteria:

* Patients with distant metastasis.
* Patients who are pregnant or breastfeeding.
* Patients with diffuse (>1 quadrant or >5 cm) suspicious microcalcifications.
* Prior radiation therapy to the ipsilateral or contralateral breast or thorax.
* Histological evidence of lymphovascular invasion (LVI). Cases termed focally suspicious for LVI but where no definitive LVI is found are eligible.
* Histologic evidence of EIC, defined as the presence of intraductal carcinoma both within the primary infiltrating ductal tumor (comprising at least 25% of the tumor area) and intraductal carcinoma present clearly beyond the edges of the invasive tumor, or as a predominantly intraductal tumor with one or more areas of focal invasion.
* Patients are not required to undergo BRCA1 and BRCA2 or other genetic mutation tests in order to enroll on the study. However, in the event a patient is tested and is found to be a mutation carrier, she would be excluded from the study. It would be an extremely rare/unlikely scenario for patients to be discovered BRCA positive after the completion of PBI, as all patients with risk factors for BRCA mutations (positive family history, Ashkenazi Jewish descent, ER-/PR-/her2-neu negative receptor status) are usually tested prior to radiation. Should such a situation exist, these patients will not receive additional RT and the patient will be replaced in the trial.
* History of cosmetic or reconstructive breast surgery.
* Psychiatric illness that would prevent the patient from giving informed consent.
* Patients for whom the delivery of PBI is not feasible
* Medical condition such as uncontrolled infection (including HIV), uncontrolled diabetes mellitus, or connective tissue diseases (lupus, systemic sclerosis, or other collagen vascular diseases) that, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient.
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have "currently active" malignancies if they have completed therapy and are considered by their physicians to be at <5% risk of relapse within 3 years.
* Patients who are already enrolled in or planning to enroll in other adjuvant systemic therapy protocols for both non-invasive or invasive breast cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2010-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of PBI-directed external-beam radiation therapy | Two weeks
  In selected stages 0 and I female breast cancer patients utilizing 40 Gy in ten daily fractions for two weeks.

SECONDARY OUTCOMES:
To evaluate local control rates | 1 year
  (local control for patients with DCIS will be analyzed separately from those patients with invasive cancer)
To evaluate distant control rates | 1 year
To evaluate breast cosmesis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Simon Powell, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering at Basking Ridge (Follow-up Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Follow-up Only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Follow-up Only), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk (Follow-up Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Follow-up Only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center (Follow-up Only), Rockville Centre, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm